CLINICAL TRIAL: NCT05850429
Title: BioDulse: The Effect of an Irish Seaweed Protein Extract on Glucose Control in Healthy Adults
Acronym: BioDulse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022_12_14_EHS
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A three arm, acute randomised, double blind crossover design feeding study will be used to establish the impact and dose response to co-ingestion of BioDulse (a protein hydrolysate from Irish seaweed) with maltodextrin on postprandial blood glucose and insulin concentrations.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): 0.6g/kg body mass maltodextrin in solution.
  Interventions: Dietary Supplement: Seaweed protein
- Low protein (Experimental): 0.6g/kg body mass maltodextrin PLUS 0.075g/kg body mass protein from Biodulse, in solution
  Interventions: Dietary Supplement: Seaweed protein
- Medium protein (Experimental): 0.6g/kg body mass maltodextrin PLUS 0.15g/kg body mass protein from Biodulse, in solution
  Interventions: Dietary Supplement: Seaweed protein

INTERVENTIONS:
Dietary Supplement: Seaweed protein — Novel protein extracted from seaweed

SUMMARY:
Co-ingesting protein with carbohydrate is an effective way to improve postprandial glucose handling. The investigators have isolated and identified a bioactive protein extracted from seaweed. The investigators aim to explore how varying doses of seaweed protein influence postprandial glycaemia and insulinaemia in a healthy population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-67

Exclusion Criteria:

* Terminal disease
* Past medical history of vascular disease, cancer, diabetes, neurological, kidney, pulmonary, digestive (Coeliac disease), thyroidal disease, cognitive impairment;
* Exclusively receiving enteral or parenteral nutrition,
* Any conditions/anomalies that are contraindications to bioelectrical impedance analysis as per institutional risk assessment and SOP.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose area under the curve (AUC) | 120 min
  Integrated area under curve of blood glucose concentration (measured as mmol/L) over 120min

SECONDARY OUTCOMES:
Timecourse of blood glucose concentration | 0, 15, 30, 45, 60, 90, 120 min
  Timecourse of blood glucose concentration (measured as mmol/L)
Postprandial serum insulin area under the curve (AUC) | 120 min
  Integrated area under curve of blood glucose concentration (measured as mU/L) over 120min
Postprandial serum insulin concentration | 0, 15, 30, 45, 60, 90, 120 min
  Timecourse of serum insulin concentration (measured as mU/L)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Carson, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with researchers outside of those named on the institutional ethics application form.